CLINICAL TRIAL: NCT05133843
Title: Complete Functional Assessment of Intermediate Coronary Artery Stenosis Before and After Transcatheter Aortic Valve Implantation (TAVI) in Patients With Severe Symptomatic Aortic Valve Stenosis
Acronym: CHOICE-FR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0125
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Stenosis; Transcatheter Aortic Valve Implantation
Keywords: Coronary Artery Stenosis; transcatheter aortic valve implantation; coronary physiology; coronary blood flow; coronary microcirculatory function; non-invasive CT-FFR; fractional flow reserve; resting full cycle ratio
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective, single center, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary physiology (Other): Assession of complete coronary physiology in TAVI candidates with intermediate coronary artery stenosis before and 6 months after TAVI.
  Interventions: Procedure: Assession of complete coronary physiology

INTERVENTIONS:
Procedure: Assession of complete coronary physiology — Assession of complete coronary physiology in TAVI candidates with intermediate coronary artery stenosis before and 6 months after TAVI.
  Other Names: FFR, RFR, CFR, IMR, and CT-FFR

SUMMARY:
The purpose of the current study is to assess complete coronary physiology (FFR, RFR, CFR, IMR, and CT-FFR) in TAVI candidates with intermediate coronary artery stenosis before and 6 months after TAVI. This aims to determine how TAVI affects coronary blood flow and coronary microcirculatory function after longer-term follow-up, and how these effects influence FFR and RFR values. In addition, it is aimed to correlate invasive functional testing (FFR and RFR) with non-invasive CT-FFR before and 6 months after TAVI.

DETAILED DESCRIPTION:
Prospective, single center, open-label study to

1. compare coronary flow reserve (CFR), index of microvascular resistance (IMR), fractional flow reserve (FFR) and resting full cycle ratio (RFR) values before TAVI and 6 months after TAVI
2. correlate testing of microcirculatory function (IMR) with measurements of functional testing (FFR and RFR) before and six months after TAVI
3. correlate functional testing (FFR and RFR) with computed tomography (CT) derived fractional flow reserve (CT-FFR) before and six months after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
* Severe symptomatic aortic stenosis with indication for TAVI according to current guidelines deemed by the Heart Team
* Patients who have undergone coronary CT angiography before TAVI in which CAD could not be ruled out
* CAD in one or more native major epicardial vessels or their branches by coronary angiogram with visually assessed coronary stenosis, in which the physiological severity of the lesion is in question (typically 40-90% diameter stenosis).
* Eligible for invasive coronary angiography and functional assessment (FFR, RFR, CFR and IMR)
* Eligible for coronary CT-angiography and functional assessment (CT-FFR)

Exclusion Criteria:

* Patients whose CT-angiography was determined to be non-diagnostic/unreadable during its evaluation
* Previous coronary artery bypass grafting with patent grafts to the interrogated vessel
* Patients with severe lesions with a diameter stenosis ≥ 90%, flow-limiting lesions, or a significant left main coronary artery stenosis
* Critical coronary artery disease deemed by the Heart Team to require immediate revascularization
* Contraindication to adenosine (e.g. bronchial asthma)
* Chronic renal impairment with severe reduction of glomerular filtration rate (eGFR <30 ml/min)
* Presence of cardiogenic shock
* Participation in another interventional study involving the left heart or coronary arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of CFR, IMR, FFR and RFR values before TAVI and 6 months after TAVI | 6 Months
  Comparison of coronary flow reserve, index of microvascular resistance, fractional flow reserve and resting full cycle ratio.
  The variation in correlation between CT-FFR and IMR, FFR or RFR before and after TAVI will be estimated using a General Linear Model (GLM) with an interaction between the independent variable (IMR, FFR, RFR) and the time period (before or after TAVI).

SECONDARY OUTCOMES:
Diagnostic accuracy by considering FFR values of >0.80 as normal | 6 Months
  diagnostic accuracy (sensitivity, specificity, positive predictive value [PPV] and negative predictive value [NPV]) of CT-FFR for the detection of significant coronary stenosis before and 6 months after TAVI by considering FFR values of >0.80 as normal
Diagnostic accuracy by considering RFR values of >0.89 as normal | 6 Months
  diagnostic accuracy (sensitivity, specificity, positive predictive value [PPV] and negative predictive value [NPV]) of CT-FFR for the detection of significant coronary stenosis before and 6 months after TAVI by considering RFR values of >0.89 as normal

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Majunke, Dr., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology; Robin Gohmann, Dr., Principal Investigator — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology; Mohamed Abdel-Wahab, Prof. Dr., Principal Investigator — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology
Locations (1):
- Heart Center Leipzig at University of Leipzig Department of Internal Medicine/Cardiology, Leipzig, Germany